CLINICAL TRIAL: NCT01089933
Title: Efficacy of Thoracic Paravertebral Block in Reducing Chronic Pain and Disability After Breast Cancer Surgery With Axillary Lymph Node Dissection
Brief Title: Reducing Pain and Disability After Breast Cancer Surgery
Acronym: RELIeF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006711-01
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Chronic Pain
Keywords: Anesthesia; Local Anesthetics; Analgesia; Quality of life; Paravertebral blocks; Arm morbidity
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Agnosia | interventions — Nerve Block; Anesthetics, Local; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic PVB + multimodal anesthesia (Experimental): Thoracic PVB + multimodal anesthesia
  Interventions: Procedure: Thoracic Paravertebral Block (TPVB)
- Local anesthetic + multi-modal analgesia (Active Comparator): Local anesthetic + multi-modal analgesia
  Interventions: Procedure: Local Anesthetic

INTERVENTIONS:
Procedure: Thoracic Paravertebral Block (TPVB) — The middle of the spinous process above the nerve to be blocked is located and the overlying skin marked 2.5 centimeters lateral to this. Subcutaneous lidocaine is injected and a 22 G Tuohy tipped 8 cm needle is inserted at this level and advanced to identify the transverse process. The needle is then moved caudad off the transverse process and inserted a centimeter into the paravertebral space. Five mls of 0.5% ropivacaine with 1:200,000 epinephrine is injected at each paravertebral space. Blocks adjacent to the C7-T5 spinous processes are performed. For patients randomized to the LA group: The patients are identically positioned, sedated and identical landmarks are used to perform sham paravertebral blocks via a subcutaneous saline injection of 0.5mL with a 25G needle at each level.
  Other Names: Regional analgesia; neural blockade
  Arms: Thoracic PVB + multimodal anesthesia
Procedure: Local Anesthetic — At the conclusion of surgery, the surgeon will infiltrate the incision with 10 ml of saline 0.9% (TPVB group) or 0.5% ropivacaine (LA group). An axillary drain will be placed. After closure of the wound, 20 ml of saline 0.9% (TPVB group) or 0.5% ropivacaine (LA group) will be injected through the drain and the drain clamped for 30 minutes after injection.
  Other Names: local anesthesia
  Arms: Local anesthetic + multi-modal analgesia

SUMMARY:
The purpose of this study is to determine if the combination of thoracic paravertebral block and multimodal analgesia will decrease chronic pain and arm morbidity in patients undergoing breast cancer surgery with lymph node dissection as compared to patients receiving local anesthesia with multimodal analgesia.

DETAILED DESCRIPTION:
Sixty percent of breast cancer patients undergo some form of breast surgery in the treatment of the early stages of the disease. The recovery from surgery can be associated with severe disabling pain persisting beyond 12 months after surgery. Research in pain has shown that early intervention of acute pain can prevent long term chronic pain.

At The Ottawa Hospital, patients receive either paravertebral blocks or wound infiltration with local anesthetic for postoperative pain management. We would like to compare these two methods of pain control to determine an analgesic technique that will reduce acute and chronic pain, and maximally improve long-term functional recovery and patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of breast cancer
* Scheduled for elective modified radical mastectomy, simple mastectomy with SLNB, breast conserving surgery (ie lumpectomy, segmental mastectomy) with ALND or ALND alone (after positive SLNB)

Exclusion Criteria:

* American Society of Anesthesiologist (ASA) class 4 or 5
* Patients with contraindications to TPVB
* Allergy to study medications
* Chronic opioid use defined as daily consumption of greater than 20 mg of oral morphine or equivalent for >7days
* Renal insufficiency defined as a creatinine clearance <40ml/min as calculated using the Cockroft-Gault formula
* Preoperative radiation therapy
* Inability to achieve normal shoulder range of motion as defined as <100o of shoulder abduction or flexion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chiu, MD, Principal Investigator — The Ottawa Hospital / Ottawa Health Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Chiu M, Bryson GL, Lui A, Watters JM, Taljaard M, Nathan HJ. Reducing persistent postoperative pain and disability 1 year after breast cancer surgery: a randomized, controlled trial comparing thoracic paravertebral block to local anesthetic infiltration. Ann Surg Oncol. 2014 Mar;21(3):795-801. doi: 10.1245/s10434-013-3334-6. Epub 2013 Oct 29. PMID 24165901
- See also: full publication, including results — https://link.springer.com/article/10.1245/s10434-013-3334-6

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thoracic PVB + Multimodal Anesthesia | Local Anesthetic + Multi-modal Analgesia
Started | 65 | 64
Completed | 65 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thoracic PVB + Multimodal Anesthesia | Local Anesthetic + Multi-modal Analgesia | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 64 | 129
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — survey was done to collect participant age
  years | 54 (10.8) | 56 (10.6) | 55 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 64 | 129
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 65 | 64 | 129

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Individuals Reporting Chronic Postoperative Pain 12 Months Following Breast Cancer Surgery With Lymph Node Dissection.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic PVB + Multimodal Anesthesia | Local Anesthetic + Multi-modal Analgesia
Number analyzed (Participants) | 65 | 64
Participants | 5 | 4

2. Secondary Outcome: Arm Morbidity, Shoulder Range of Motion, Quality of Analgesia, Arm Lymphedema, Time to Meet Discharge Criteria, Quality of Recovery, Quality of Life, Incidence of Postoperative Side Effects.
Description: Brief Pain Inventory (BPI); Flexion, extension, abduction, internal, and external rotation of the shoulder; Constant score; Quality of life was assessed using the FACTB4 and the SF-12 Health Survey (SF12); Details of the surgery, chemotherapy, and/or radiation therapy were recorded
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Arm/Group | Thoracic PVB + Multimodal Anesthesia | Local Anesthetic + Multi-modal Analgesia
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/64
Other Adverse Events (participants affected / at risk) | 0/65 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No